CLINICAL TRIAL: NCT04442022
Title: A Phase 2/3, Multicenter Randomized Study of Rituximab-Gemcitabine-Dexamethasone-Platinum (R-GDP) With or Without Selinexor in Patients With Relapsed/Refractory Diffuse Large B-cell Lymphoma (RR DLBCL)
Brief Title: A Study of Rituximab-Gemcitabine-Dexamethasone-Platinum (R-GDP) With or Without Selinexor in Patients With Relapsed/Refractory Diffuse Large B-cell Lymphoma
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: XPORT-DLBCL-030; 2020-000605-84 (EudraCT Number)
Record Dates: First submitted 2020-06-10; First posted 2020-06-22 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Relapsed/Refractory Diffuse Large B-cell Lymphoma
Keywords: Relapsed/Refractory DLBCL; Rituximab-Gemcitabine-Dexamethasone-Platinum (R-GDP); Selinexor; Karyopharm; KCP-330; XPOVIO; DLBCL; XPORT-DLBCL-030; R-GDP
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence | interventions — selinexor; Combined Modality Therapy; Rituximab; Gemcitabine; Dexamethasone; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Phase 2 Portion of the Study: open label; Phase 3 Portion of the Study: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Phase 2: Selinexor 40 mg + R-GDP (Experimental): Patients with RR DLBCL will receive combination therapy of selinexor 40 mg orally at Day 1 and Day 8 of each 21-day cycle for up to 6 cycles in combination with R-GDP followed by single-agent continuous therapy with selinexor 60 mg orally once weekly (QW) for each 28-day cycle until progressive disease (PD) or unacceptable toxicity.
  Interventions: Drug: Selinexor (combination therapy); Drug: Rituximab (combination therapy); Drug: Gemcitabine (combination therapy); Drug: Dexamethasone (combination therapy); Drug: Cisplatin (combination therapy); Drug: Selinexor (continuous therapy)
- Phase 2: Selinexor 60 mg + R-GDP (Experimental): Patients with RR DLBCL will receive combination therapy of selinexor 60 mg orally at Day 1 and Day 8 of each 21-day cycle for up to 6 cycles in combination with R-GDP followed by single-agent continuous therapy with selinexor 60 mg orally QW for each 28-day cycle until PD or unacceptable toxicity.
  Interventions: Drug: Selinexor (combination therapy); Drug: Rituximab (combination therapy); Drug: Gemcitabine (combination therapy); Drug: Dexamethasone (combination therapy); Drug: Cisplatin (combination therapy); Drug: Selinexor (continuous therapy)
- Phase 2: R-GDP (Active Comparator): Patients with RR DLBCL will receive R-GDP on specified days (Days 1, 2, 3, 4, and 8) for each 21-day cycle for up to 6 cycles.
  Interventions: Drug: Rituximab (combination therapy); Drug: Gemcitabine (combination therapy); Drug: Dexamethasone (combination therapy); Drug: Cisplatin (combination therapy)
- Phase 3: Selinexor (Selected Dose) + R-GDP followed by Selinexor 60 mg (Experimental): Patients with RR DLBCL will receive combination therapy of selinexor (selected dose from Phase 2) at Day 1 and Day 8 of each 21-day cycle for up to 6 cycles in combination with R-GDP followed by selinexor 60 mg orally QW for each 28-day cycle until PD or unacceptable toxicity.
  Interventions: Drug: Selinexor (combination therapy); Drug: Rituximab (combination therapy); Drug: Gemcitabine (combination therapy); Drug: Dexamethasone (combination therapy); Drug: Cisplatin (combination therapy); Drug: Selinexor (continuous therapy)
- Phase 3: Selinexor (Selected Dose) + R-GDP followed by Placebo (Experimental): Patients with RR DLBCL will receive combination therapy of selinexor (selected dose from Phase 2) at Day 1 and Day 8 of each 21-day cycle for up to 6 cycles in combination with R-GDP followed by matching placebo for selinexor orally QW for each 28-day cycle until PD or unacceptable toxicity.
  Interventions: Drug: Selinexor (combination therapy); Drug: Rituximab (combination therapy); Drug: Gemcitabine (combination therapy); Drug: Dexamethasone (combination therapy); Drug: Cisplatin (combination therapy); Drug: Placebo matching for Selinexor (continuous therapy)
- Phase 3: Placebo + R-GDP followed by Placebo (Placebo Comparator): Patients with RR DLBCL will receive combination therapy of placebo matching for selinexor (selected dose from Phase 2) at Day 1 and Day 8 of each 21-day cycle for up to 6 cycles in combination with R-GDP followed by matching placebo for selinexor orally QW for each 28-day cycle until PD or unacceptable toxicity.
  Interventions: Drug: Placebo matching for Selinexor (combination therapy); Drug: Rituximab (combination therapy); Drug: Gemcitabine (combination therapy); Drug: Dexamethasone (combination therapy); Drug: Cisplatin (combination therapy); Drug: Placebo matching for Selinexor (continuous therapy)

INTERVENTIONS:
Drug: Selinexor (combination therapy) — Dose: 40 mg on Days 1 and 8 of each 21-day cycle for up to 6 cycles; Route of administration: oral
  Arms: Phase 2: Selinexor 40 mg + R-GDP
Drug: Selinexor (combination therapy) — Dose: 60 mg on Days 1 and 8 of each 21-day cycle for up to 6 cycles; Route of administration: oral
  Arms: Phase 2: Selinexor 60 mg + R-GDP
Drug: Selinexor (combination therapy) — Dose: Selected dose of selinexor (from Phase 2) on Days 1 and 8 of each 21-day cycle for up to 6 cycles; Route of administration: oral
  Arms: Phase 3: Selinexor (Selected Dose) + R-GDP followed by Placebo; Phase 3: Selinexor (Selected Dose) + R-GDP followed by Selinexor 60 mg
Drug: Placebo matching for Selinexor (combination therapy) — Dose: Placebo matching for selected dose of selinexor (from Phase 2) on Days 1 and 8 of each 21-day cycle for up to 6 cycles; Route of administration: oral
  Arms: Phase 3: Placebo + R-GDP followed by Placebo
Drug: Rituximab (combination therapy) — Dose: 375 milligram per meter square (mg/m^2) on Day 1; Route of administration: intravenous (IV)
  Arms: Phase 2: Selinexor 40 mg + R-GDP
Drug: Rituximab (combination therapy) — Dose: 375 mg/m^2 on Day 1; Route of administration: IV
  Arms: Phase 2: R-GDP; Phase 2: Selinexor 60 mg + R-GDP; Phase 3: Placebo + R-GDP followed by Placebo; Phase 3: Selinexor (Selected Dose) + R-GDP followed by Placebo; Phase 3: Selinexor (Selected Dose) + R-GDP followed by Selinexor 60 mg
Drug: Gemcitabine (combination therapy) — Dose: 1000 mg/m^2 on Days 1 and 8; Route of administration: IV
Drug: Dexamethasone (combination therapy) — Dose: 40 mg (20 mg if patient is more than 70 years old) on Days 1, 2, 3, and 4; Route of administration: oral or IV
Drug: Cisplatin (combination therapy) — Dose: 75 mg/m^2 on Day 1; Route of administration: IV
Drug: Selinexor (continuous therapy) — Dose: 60 mg QW for each 28-day cycle until PD; Route of administration: oral
  Arms: Phase 2: Selinexor 40 mg + R-GDP; Phase 2: Selinexor 60 mg + R-GDP; Phase 3: Selinexor (Selected Dose) + R-GDP followed by Selinexor 60 mg
Drug: Placebo matching for Selinexor (continuous therapy) — Dose: Placebo matching for 60 mg selinexor QW for each 28-day cycle until PD; Route of administration: oral
  Arms: Phase 3: Placebo + R-GDP followed by Placebo; Phase 3: Selinexor (Selected Dose) + R-GDP followed by Placebo

SUMMARY:
The purpose of this Phase 2/3 study is to evaluate efficacy and safety of the combination of selinexor and R-GDP (SR-GDP) in patients with RR DLBCL who are not intended to receive hematopoetic stem cell transplantation (HSCT) or chimeric antigen receptor T cell (CAR-T) therapy. This study consists of 3 arms each in Phase 2 and 3. Phase 2 portion of the study will assess the two doses of selinexor (40 milligram [mg] or 60 mg) in combination with R-GDP, for up to 6 cycles (21-day per cycle), followed by 60 mg selinexor single agent continuous therapy for those who have reached a partial or complete response. Phase 3 portion of the study will evaluate the selected dose of SR-GDP (identified in Phase 2) versus standard R-GDP + matching placebo, for up to 6 cycles (21-day per cycle), followed by placebo or 60 mg selinexor single agent continuous therapy for those who have reached partial or complete response.

ELIGIBILITY:
Inclusion Criteria:

* Have pathologically confirmed de novo DLBCL or DLBCL transformed from previously diagnosed indolent lymphoma (e.g., follicular lymphoma). Patient with high-grade lymphoma with c-MYC, Bcl2 and/or Bcl6 rearrangements are eligible (only for Phase 2). (Documentation to be provided).
* Have received at least 1 but no more than 3 prior lines of systemic therapy for the treatment of DLBCL with relapsed or refractory disease following their most recent regimen.

  * Salvage chemoimmunotherapy followed by stem cell transplantation will be considered as 1 line of systemic therapy.
  * Maintenance therapy will not be counted as a separate line of systemic therapy.
  * Radiation with curative intent for localized DLBCL will not be counted as 1 line of systemic therapy.
* Positron emission tomography (PET) positive measurable disease with at least 1 node having the longest diameter (LDi) greater than (>) 1.5 centimeter (cm) or 1 extranodal lesion with LDi >1 cm (per the Lugano Criteria 2014). The Deauville 5-point scale (D5PS) score assessed on the FDG PET/CT should be between 3 to 5.
* Not intended for HSCT or CAR-T cell therapy based on objective clinical criteria determined by the treating physician. Patients who cannot receive HSCT due to active disease are allowed on study (up to approximately 15 percent [%] of patients enrolled in each Phase). Documentation on lack of intention to proceed to receive HSCT or CAR-T therapy must be provided by the treating physician.
* Adequate bone marrow function at screening, defined as:

  * Absolute neutrophil count (ANC) ≥1*10^9 per liter (/L).
  * Platelet count ≥100*10^9/L (without platelet transfusion less than [<] 14 days prior to Cycle 1 Day 1 [C1D1]).
  * Hemoglobin ≥8.5 gram per deciliter (g/dL) (without red blood cell transfusion <14 days prior to C1D1).
* Circulating lymphocytes less than or equal to (≤) 50*10^9/L.
* Adequate liver and kidney function, defined as:

  * Aspartate transaminase (AST) or alanine transaminase (ALT) ≤2.5*upper limit of normal (ULN), or ≤5*ULN in cases with known lymphoma involvement in the liver.
  * Serum total bilirubin ≤2*ULN, or ≤5*ULN if due to Gilbert syndrome or in cases with known lymphoma involvement in the liver.
  * Calculated creatinine clearance (CrCl) ≥30 milliliter per minute (mL/min) based on Cockcroft-Gault formula.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
* An estimated life expectancy of >3 months at Screening.
* Patients with primary refractory DLBCL defined as no response or relapse within 6 months after ending first-line treatment, will be allowed in the study.
* Agree to highly effective contraception during the duration of the study with contraception use continuing for 12 months after the last dose of study treatment
* Female patients of childbearing potential must have a negative serum pregnancy test at Screening and agree to use highly effective methods of contraception throughout the study and for 12 months following the last dose of study treatment (except patients with Non-Childbearing potential: Age >50 years and naturally amenorrhoeic for >1 year, or previous bilateral salpingo-oophorectomy, or hysterectomy).
* Male patients who are sexually active must use highly effective methods of contraception throughout the study and for 12 months following the last dose of study treatment. Male patients must agree not to donate sperm during the study treatment period and for 12 months following the last dose of study treatment.

Exclusion Criteria:

* DLBCL with mucosa-associated lymphoid tissue (MALT) lymphoma, composite lymphoma (Hodgkin's lymphoma + non-Hodgkin's lymphoma [NHL]), DLBCL transformed from diseases other than indolent NHL; primary mediastinal (thymic) large B-cell lymphoma (PMBL); T-cell rich large B-cell lymphoma.
* Previous treatment with selinexor or other XPO1 inhibitors.
* Contraindication to any drug contained in the combination therapy regimen (SR-GDP).
* Known active central nervous system or meningeal involvement by DLBCL at time of Screening.
* Use of any standard or experimental anti-DLBCL therapy (including nonpalliative radiation, chemotherapy, immunotherapy, radio-immunotherapy, or any other anticancer therapy) <21 days prior to C1D1 (prednisone <30 mg or equivalent is permitted; palliative radiation is permitted only if on non-target lesions).
* Any AE, by C1D1, which has not recovered to Grade ≤1 (Common Terminology Criteria for Adverse Events [CTCAE], v.5.0), or returned to baseline, related to the previous DLBCL therapy, except hematological abnormalities (as specified in the inclusion criteria) and alopecia.
* Major surgery <14 days of Cycle 1 Day 1.
* Hematopoietic stem cell transplantation/CAR-T therapy as follows:

  * Autologous stem cell transplant (SCT) <100 days or allogeneic-SCT <180 days prior to C1D1
  * Active graft-versus-host disease (GVHD) after allogeneic SCT (or cannot discontinue GVHD treatment or prophylaxis)
  * CAR-T cell infusion <90 days prior to Cycle 1
* Neuropathy Grade ≥2 (CTCAE, v.5.0).
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the Investigator's opinion, could compromise the patient's safety, or being compliant with the study procedures.
* Uncontrolled (i.e., clinically unstable) infection requiring parenteral antibiotics, antivirals, or antifungals within 7 days prior to first dose of study treatment; however, prophylactic use of these agents is acceptable (including parenteral).
* Patient with active hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) infections:

  * Patient with active HBV are allowed if antiviral therapy for hepatitis B has been given for >8 weeks and viral load is <100 International units (IU)/mL prior to first dose of study treatment.
  * Patients with known history of HCV or found to be HCV antibody positive on screening, are allowed if there is documentation of negative viral load per institutional standard.
  * Patients with HIV are allowed if they have a negative viral load per institutional standard, and no history of acquired immune deficiency syndrome (AIDS)-defining opportunistic infections in the last year.
* Inability to swallow tablets, malabsorption syndrome, or any other gastrointestinal (GI) disease or dysfunction that could interfere with absorption of study treatment.
* Breastfeeding or pregnant women.
* Inability or unwillingness to sign an informed consent form (ICF).
* In the opinion of the Investigator, patient who are significantly below their ideal body weight.
* Patients who received a live attenuated vaccine within prior 28 days of the first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Estimated)
Dates: Start 2020-09-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Phase 2: Overall Response Rate (ORR): Based on Lugano Criteria 2014 | From date of initial randomization to the date of disease progression or initiating a new DLBCL treatment (maximum of 5 years from randomization)
Phase 3: Progression-free Survival (PFS): Based on Lugano Criteria 2014 | From date of initial randomization to the date of disease progression or death (maximum of 5 years from randomization)

SECONDARY OUTCOMES:
Phase 2: Progression-free Survival: Based on Lugano Criteria 2014 | From date of initial randomization to the date of disease progression or death (maximum of 5 years from randomization)
Phase 2: Overall Survival (OS) | From date of initial randomization until death (maximum of 5 years from randomization)
Phase 3: Overall Response Rate: Based on Lugano Criteria 2014 | From date of initial randomization to the date of disease progression or initiating a new DLBCL treatment (maximum of 5 years from randomization)
Phase 3: Overall Survival | From date of initial randomization until death (maximum of 5 years from randomization)
Phase 2: Overall Response Rate at the End of Combination Therapy (ORR-EoC): Based on Lugano Criteria 2014 | From C1D1 (Cycles 1 up to 6; 21 days per cycle) up to 28 days after EoC therapy
Phase 2: Overall Response Rate at the End of Combination Therapy: Based on Modified Lugano Criteria | From C1D1 (Cycles 1 up to 6; 21 days per cycle) up to 28 days after EoC therapy
Phase 2: Duration of Response (DOR): Based on Lugano Criteria 2014 | From time of first response until disease progression or death (maximum of 5 years from randomization)
Phase 2: Number of Patients with Adverse Events (AEs) | Up to 30 days after last dose of study drug (maximum of 5 years from randomization)
Phase 3: Overall Response Rate at the End of Combination Therapy: Based on Lugano Criteria 2014 | From C1D1 (Cycles 1 up to 6; 21 days per cycle) up to 28 days after EoC therapy
Phase 3: Overall Response Rate at the End of Combination Therapy: Based on Modified Lugano Criteria | From C1D1 (Cycles 1 up to 6; 21 days per cycle) up to 28 days after EoC therapy
Phase 3: Duration of Response: Based on Lugano Criteria 2014 | From time of first response until disease progression or death (maximum of 5 years from randomization)
Phase 3: Progression-free Survival: Based on Modified Lugano Criteria | From date of initial randomization to the date of disease progression or death (maximum of 5 years from randomization)
Phase 3: Number of Patients with Adverse Events | Up to 30 days after last dose of study drug (maximum of 5 years from randomization)

CONTACTS AND LOCATIONS:
Locations (57):
- United States (19):
  - Ironwood Physicians P.C. dba Ironwood Cancer and Research Centers, Chandler, Arizona
  - Arizona Oncology Associates, Tucson, Arizona
  - The Oncology Institute (TOI) Clinical Research, Cerritos, California
  - Investigative Clinical Research of Indiana, LLC, Indianapolis, Indiana
  - Norton Cancer Institute, St. Matthews, Louisville, Kentucky
  - Tulane Cancer Center, New Orleans, Louisiana
  - University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - Stony Brook, Stony Brook, New York
  - Gabrail Cancer Center Research LLC, Canton, Ohio
  - Texas Oncology - Medical City Dallas, Dallas, Texas
  - Texas Oncology - Presbyterian Dallas Cancer Center, Dallas, Texas
  - Texas Oncology - Sammons, Dallas, Texas
  - Texas Oncology - Fort Worth, Fort Worth, Texas
  - Texas Oncology - Plano East, Plano, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - The University of Texas Health Science Center at Tyler DBA UT Health East Texas HOPE Cancer Center, Tyler, Texas
  - Providence Regional Cancer Partnership, Everett, Washington
- Austria (3):
  - Kepler Universitaetskrankenhaus Med Campu III - Onkologie, Linz, Austria
  - University of Vienna, Medical Clinic I, Hematology, Vienna, Austria
  - Hospital Hietzing, Vienna, Austria
- China (6):
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Ruijin Hospital Affiliated to The Shanghai Jiao Tong University Medical School, Huangpu, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Xuhui, Shanghai Municipality
  - Huaxi Hospital Sichuan University, Chengdu, Sichuan
  - The first affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
- Israel (8):
  - Assuta Ashdod Medical Center, Ashdod
  - Soroka Medical Center, Beersheba
  - Rambam health care campus (Department of Hematology & Bone Marrow Transplantation), Haifa
  - Wolfson Medical Center, Holon
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Assuta medical centers - Ramat Hachayal, Tel Aviv
  - Sourasky Medical Center, Tel Aviv
- Italy (9):
  - AOU Ospedali Riuniti-Università Politecnica delle Marche Clinica di Ematologia, Ancona, Ancona
  - AOU Policlinico S.Orsola Malpighi di Bologna, University of Bologna, Bologna, Bologna
  - UOC Ematologia ad Indirizzo Oncologico, AORN "Sant'Anna e San Sebastiano", Caserta, Caserta
  - National Cancer Institute, Naples, Napoli
  - AOU Maggiore della Carità SCDU Ematologia, Novara, Novara
  - DIP. Oncologia- Ematologia, UOSD Centro Diagnosie TerapiaDei Linfomi, Pescara, Pescara
  - Fondatione Policlinico Universitario A. Gemelli, Rome, Rome
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello, Palermo, Sicily
  - AOU City of Health and Science of Turin, Turin, Torino
- Poland (7):
  - Pratia MCM Krakow, Krakow, Lesser
  - Szpitale pomorskie gdynia dept of haematology, Gdynia, Pomeranian Voivodeship
  - Klinika Hematologii, Nowotworów Krwi i Transplantacji Szpiku Uniwersytecki Szpital Kliniczny im. Jana Mikulicza - Radeckiego we Wrocławiu, Wroclaw, Radeckiego
  - Pratia Onkologia Katowice, Katowice, Silesian Voivodeship
  - CM Pratia Poznań, Skorzewo, Wielkopolska
  - Institute of Hematology and Transfusion Medicine, Warsaw
  - Department of Lymphoid Malignancies, Maria Sklodowska-Curie National Research Institute of Oncology, Warsaw
- Spain (5):
  - Institut català d'oncologia-hospital germans trias i pujol, Badalona, Barcelona
  - Hospital Vall Hebron, Barcelona, Barcelona
  - Institut Catala D'oncolocia, Barcelona, Barcelona
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Virgen del Rocío, Seville, Seville

IPD SHARING:
Plan to Share IPD: Undecided